CLINICAL TRIAL: NCT06630715
Title: Efficacy Of Upadacitinib In Psoriatic Arthritis And Comparison To Rheumatoid Arthritis. OPTimising IMAging For The Use In The Follow-Up Of Arthritis: The OPTIMA Study
Brief Title: Efficacy Of Upadacitinib In Psoriatic Arthritis And Comparison To Rheumatoid Arthritis.
Acronym: OPTIMA
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: OPTIMA (L4182)
Record Dates: First submitted 2024-09-25; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis (RA; Psoriatic Arthritis (PsA
Keywords: rheumathoid Arthritis; Psoriatic Arthritis; Ultrasound; MRI; Upadacitinib; Dactylitis; Enthesitis; Synovitis; sacroiliitis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic; Salivary Gland Adenoma, Pleomorphic; Synovitis; Sacroiliitis | interventions — upadacitinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis: Patients diagnosed with RA according to the ACR/EULAR 2010 classification criteria with active disease starting Upadacitinib
  Interventions: Drug: Upadacitinib 15 MG [Rinvoq]
- Psoriatic Arthritis: Patients diagnosed with peripheral Psoriatic Arthritis according to the CASPAR criteria or with axial Psoriatic Arthritis according to ASAS criteria with active disease starting Upadacitinib
  Interventions: Drug: Upadacitinib 15 MG [Rinvoq]

INTERVENTIONS:
Drug: Upadacitinib 15 MG [Rinvoq] — 15 mg/ day

SUMMARY:
The general objective of the OPTIMA study is to assess the time course and interrelationship of imaging (ultrasound and magnetic resonance imaging), clinical, laboratory, and Patient Reported Outcome variables in patients with active Psoriatic Arthritis (any subset) and Rheumatoid Arthritis starting therapy with a Jak-Inhibitor (Upadacitinib), during the first 6 months of follow-up.

Participants will be evaluated at the start of therapy with upadacitinib and during the follow-up visits at 2 weeks, 1, 3, and 6 months post-treatment initiation. At each visit (with the exception of the 2-weeks visit), data relating to the clinical evaluation, laboratory tests, and ultrasound of the affected joints will be collected according to standard clinical practice; questionnaires on disease activity will also be completed. In the case of axial involvement, a magnetic resonance imaging will be performed at baseline and after 6 months of therapy, only if required by the standard of care.

DETAILED DESCRIPTION:
This is a multicentric prospective observational study in which consecutive patients diagnosed with Psoriatic Arthritis (any subset) and Rheumatoid Arthritis, that according to clinicians' evaluation should be treated with Upadacitinib therapy, will be recruited from the outpatient clinic of the Rheumatology Department of the centers included in the study.

The investigators will enroll consecutive patients with Psoriatic Arthritis and Rheumatoid Arthritis with active disease and fulfilling the inclusion and exclusion criteria, from the outpatient clinic of the Rheumatology Units of the participating centers. Written informed consent will be obtained prior to the beginning of the study. All patients, in line with clinical routine practice, will undergo a standard clinical, laboratory, and imaging assessment in order to define the disease activity according to standardized disease activity indexes, at baseline and during the first 3 follow-up visits. For patients starting new treatments for Psoriatic Arthritis and Rheumatoid Arthritis, the follow-up visits are generally scheduled after 1 month (± 1 week), 3 months (± 2 weeks), and 6 months (± 4 weeks) post-treatment initiation, in accordance with international guidelines and local protocols. In case of suspicion of axial involvement, an MRI of the sacroiliac joints will be performed at baseline and, in case of positivity, will be repeated after 6 months (±1 month) in order to assess disease activity at the spine and the treatment efficacy. Regarding the Patient Reported Outcome, the investigators will assess these during the scheduled visits, and two weeks after the initiation of treatment to evaluate earlier pain and functional improvement. The Patient Reported Outcome assessment at two weeks will be administered in a paper form to participants during the baseline visit, and subsequently participants will return these during the first follow-up visit. The data for the study will be retrieved from the medical records of participants and recorded into an appositely created electronic case report form.

ELIGIBILITY:
The inclusion criteria for Psoriatic Arthritis patients are:

1. Patients diagnosed with peripheral Psoriatic Arthritis according to the CASPAR criteria or with axial Psoriatic Arthritis according to ASAS criteria and with at least one of the following:

   1. With active peripheral Psoriatic Arthritis regarding ongoing therapy in one of the following sites: MCP joints 1-5, proximal interphalangeal (PIP) joints of hands 1-5, distal interphalangeal (DIP) joints of hands 2-5, wrists, elbows, knees and ankles/heels and feet, according to any of the following criteria:

      I) DAPSA ≥ 15 and joint inflammation according to the Global OMERACT-EULAR US scoring for synovitis and power Doppler (GLOESS) with a grade at patient level >3,2

      II) With a clinical enthesitis and an active enthesitis (positive power Doppler of any grade), in the clinical symptomatic site, according to the OMERACT US definitions

      III) With active dactylitis (clinical diagnosis made by the physician at the time of baseline visit) and a positive US dactylitis according to the DACTylitis glObal Sonographic (DACTOS) score >3

      IV) DAPSA ≥ 15 and tenosynovitis according to the OMERACT US scoring system for tenosynovitis with a grade >1
   2. With active axial PsA regarding ongoing therapy (ASDAS ≥ 2.1) and active sacroiliitis according to the ASAS MRI definitions
2. Who are eligible according to the current guidelines/regulations to start treatment with UPA and present a favorable risk/benefit profile according to the clinician's opinion for such treatment.
3. Aged older than 18 years.
4. Able to provide informed consent, according to requirements of local IRB/ethics committee.

The inclusion criteria for Rheumatoid Arthritis patients are:

1. Patients diagnosed with RA according to the ACR/EULAR 2010 classification criteria
2. With active Rheumatoid Arthritis according to the following criteria: DAS28-PCR >3.2, and the presence of at least one US finding of the following:

   1. Joint inflammation at hands and wrists according to the Global OMERACT-EULAR (GLOESS) US scoring for synovitis and power Doppler with a grade at patient level >2
   2. One tenosynovitis at hands or wrists, according to the OMERACT US scoring system for tenosynovitis with a grade >1
3. Who are eligible according to the current guidelines/regulations to start treatment with Upadacitinib and present a favourable risk/benefit profile according to the clinician's opinion for such treatment.
4. Aged older than 18 years.
5. Able to provide informed consent, according to requirements of local IRB/ethics committee.

Exclusion Criteria:

1. Patients with any contraindication to Upadacitinib:

   1. women who are pregnant or breastfeeding
   2. active infection
   3. evidence of tuberculosis infection
   4. known infection with human immunodeficiency virus or hepatitis B or C
   5. patients who have current malignancy or history of malignancy in the last 5 years
   6. high cardiovascular risk
   7. high risk of venous thromboembolism
   8. patients with severe hepatic impairment
2. Patients with associated fibromyalgia syndrome according to the 2016 ACR diagnostic criteria
3. Unable to provide informed consent, according to requirements of local IRB/ethics committee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with active Psoriatic Arthritis and patients with active Rheumatoid Arthritis who will start therapy with upadacitinib
Sampling Method: Non-Probability Sample
Enrollment: 178 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Difference between US synovitis score | from baseline to 24 weeks
  Difference between US synovitis score from baseline to 24 weeks in patients with active synovitis

SECONDARY OUTCOMES:
Difference between US dactylitis score | from baseline to 24 weeks
  Difference between US dactylitis score (DACTOS) from baseline to 24 weeks in patients with active dactylitis
Difference between US tenosynovitis score | from baseline to 24 weeks
  Difference between US tenosynovitis score from baseline to 24 weeks in patients with active tenosynovitis
Difference between US enthesitis score | from baseline to 24 weeks
  Difference between US enthesitis score from baseline to 24 weeks in patients with active enthesitis
Difference between US peritendonitis score | from baseline to 24 weeks
  Difference between US peritendonitis score from baseline to 24 weeks in patients with peritendonitis
Difference between SPARCC MRI index | from baseline to 24 weeks
  Difference between SPARCC MRI index from baseline to 24 weeks in patients with active sacroiliitis in PsA
Difference between T2 mapping scores | from baseline to 24 weeks
  Difference between T2 mapping scores from baseline to 24 weeks in patients with active sacroiliitis in PsA
Difference between SJC66 | from baseline to 24 weeks
  Difference between SJC66 from baseline to 24 weeks in PsA and RA
Difference between TJC68 | from baseline to 24 weeks
  Difference between TJC68 from baseline to 24 weeks in PsA and RA
Difference between the SPARCC score | from baseline to and 24 weeks
  Difference between the SPARCC score from baseline to and 24 weeks in PsA
Difference between the dactylitis count | from baseline to 24 weeks
  Difference between the dactylitis count from baseline to and 24 weeks in PsA
Prevalence of BSA = 0 | after 24 weeks
  Prevalence of BSA = 0 after 24 weeks in PsA
Difference between CRP levels | from baseline to and 24 weeks
  Difference between CRP levels from baseline to and 24 weeks in PsA and RA
Difference between HAQ score | from baseline to and 24 weeks
  Difference between HAQ score from baseline to and 24 weeks in PsA and RA
Difference between Physician's Global Assessment of Disease Activity VAS | from baseline to and 24 weeks
  Difference between Physician's Global Assessment of Disease Activity VAS from baseline to and 24 weeks in PsA and RA
Difference between VAS pain | from baseline to and 24 weeks
  Difference between VAS pain from baseline to and 24 weeks in PsA and RA
Difference between GH-VAS | from baseline to 24 weeks
  Difference between GH-VAS from baseline to and 24 weeks in PsA and RA
Difference between ASDAS levels | from baseline to 24 weeks
  Difference between ASDAS levels from baseline to and 24 weeks in PsA
Prevalence of MDA | at 24 weeks
  Prevalence of MDA at 24 weeks in PsA
Difference between DAS28 levels | baseline and 24 weeks
  Difference between DAS28 levels at baseline and 24 weeks in PsA and RA
Time to remission | up to 2 weeks
  Time to remission in PsA and RA up to 2 weeks
Adverse events | from baseline and 24 weeks
  Adverse events from baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Filippou, MD, Principal Investigator — Università degli Studi di Milano / IRCCS Ospedale Galeazzi-Sant'Ambrogio
Locations (14):
- Italy (14):
  - Ospedale Civile di Legnano, Legnano, Milano
  - IRCCS Ospedale Humanitas, Rozzano, Milano
  - IRCCS Policlinico San Donato, San Donato, Milano
  - IRCCS Ospedale Galeazzi-Sant'Ambrogio,, Milan, Mi
  - IRCCS San Gerardo, Monza, Monza E Brianza
  - ASST Papa Giovanni XXIII, Bergamo
  - ASST Spedali Civili, Brescia
  - ASST Gaetano Pini CTO, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - ASST Fatebenefratelli-Sacco Ospedale Luigi Sacco, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - IRCCS Istituti Clinici Scientifici Maugeri, Pavia
  - ASST Settelaghi - Ospedale di Circolo di Varese, Varese

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Albano D, Bignone R, Chianca V, Cuocolo R, Messina C, Sconfienza LM, Ciccia F, Brunetti A, Midiri M, Galia M. T2 mapping of the sacroiliac joints in patients with axial spondyloarthritis. Eur J Radiol. 2020 Oct;131:109246. doi: 10.1016/j.ejrad.2020.109246. Epub 2020 Aug 29. PMID 32911127
- [Background] Maksymowych WP, Inman RD, Salonen D, Dhillon SS, Williams M, Stone M, Conner-Spady B, Palsat J, Lambert RG. Spondyloarthritis research Consortium of Canada magnetic resonance imaging index for assessment of sacroiliac joint inflammation in ankylosing spondylitis. Arthritis Rheum. 2005 Oct 15;53(5):703-9. doi: 10.1002/art.21445. PMID 16208659
- [Background] Lambert RG, Bakker PA, van der Heijde D, Weber U, Rudwaleit M, Hermann KG, Sieper J, Baraliakos X, Bennett A, Braun J, Burgos-Vargas R, Dougados M, Pedersen SJ, Jurik AG, Maksymowych WP, Marzo-Ortega H, Ostergaard M, Poddubnyy D, Reijnierse M, van den Bosch F, van der Horst-Bruinsma I, Landewe R. Defining active sacroiliitis on MRI for classification of axial spondyloarthritis: update by the ASAS MRI working group. Ann Rheum Dis. 2016 Nov;75(11):1958-1963. doi: 10.1136/annrheumdis-2015-208642. Epub 2016 Jan 14. PMID 26768408
- [Background] Sudol-Szopinska I, Jurik AG, Eshed I, Lennart J, Grainger A, Ostergaard M, Klauser A, Cotten A, Wick MC, Maas M, Miese F, Egund N, Boutry N, Rupreht M, Reijnierse M, Oei EH, Meier R, O'Connor P, Feydy A, Mascarenhas V, Plagou A, Simoni P, Platzgummer H, Rennie WJ, Mester A, Teh J, Robinson P, Guglielmi G, Astrom G, Schueller-Weiderkamm C. Recommendations of the ESSR Arthritis Subcommittee for the Use of Magnetic Resonance Imaging in Musculoskeletal Rheumatic Diseases. Semin Musculoskelet Radiol. 2015 Sep;19(4):396-411. doi: 10.1055/s-0035-1564696. Epub 2015 Nov 19. PMID 26583367
- [Background] Torp-Pedersen S, Christensen R, Szkudlarek M, Ellegaard K, D'Agostino MA, Iagnocco A, Naredo E, Balint P, Wakefield RJ, Torp-Pedersen A, Terslev L. Power and color Doppler ultrasound settings for inflammatory flow: impact on scoring of disease activity in patients with rheumatoid arthritis. Arthritis Rheumatol. 2015 Feb;67(2):386-95. doi: 10.1002/art.38940. PMID 25370843
- [Background] Moller I, Janta I, Backhaus M, Ohrndorf S, Bong DA, Martinoli C, Filippucci E, Sconfienza LM, Terslev L, Damjanov N, Hammer HB, Sudol-Szopinska I, Grassi W, Balint P, Bruyn GAW, D'Agostino MA, Hollander D, Siddle HJ, Supp G, Schmidt WA, Iagnocco A, Koski J, Kane D, Fodor D, Bruns A, Mandl P, Kaeley GS, Micu M, Ho C, Vlad V, Chavez-Lopez M, Filippou G, Ceron CE, Nestorova R, Quintero M, Wakefield R, Carmona L, Naredo E. The 2017 EULAR standardised procedures for ultrasound imaging in rheumatology. Ann Rheum Dis. 2017 Dec;76(12):1974-1979. doi: 10.1136/annrheumdis-2017-211585. Epub 2017 Aug 16. PMID 28814430
- [Background] Gutierrez M, Filippucci E, Salaffi F, Di Geso L, Grassi W. Differential diagnosis between rheumatoid arthritis and psoriatic arthritis: the value of ultrasound findings at metacarpophalangeal joints level. Ann Rheum Dis. 2011 Jun;70(6):1111-4. doi: 10.1136/ard.2010.147272. Epub 2011 Mar 15. PMID 21406459
- [Background] Moon SJ, Lee WY, Hwang JS, Hong YP, Morisky DE. Accuracy of a screening tool for medication adherence: A systematic review and meta-analysis of the Morisky Medication Adherence Scale-8. PLoS One. 2017 Nov 2;12(11):e0187139. doi: 10.1371/journal.pone.0187139. eCollection 2017. PMID 29095870
- [Background] Horta-Baas G. Patient-Reported Outcomes in Rheumatoid Arthritis: A Key Consideration for Evaluating Biosimilar Uptake? Patient Relat Outcome Meas. 2022 Mar 30;13:79-95. doi: 10.2147/PROM.S256715. eCollection 2022. PMID 35388274
- [Background] Oji V, Luger TA. The skin in psoriasis: assessment and challenges. Clin Exp Rheumatol. 2015 Sep-Oct;33(5 Suppl 93):S14-9. Epub 2015 Oct 15. PMID 26472560
- [Background] Maksymowych WP, Mallon C, Morrow S, Shojania K, Olszynski WP, Wong RL, Sampalis J, Conner-Spady B. Development and validation of the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index. Ann Rheum Dis. 2009 Jun;68(6):948-53. doi: 10.1136/ard.2007.084244. Epub 2008 Jun 4. PMID 18524792
- [Background] Duarte-Garcia A, Leung YY, Coates LC, Beaton D, Christensen R, Craig ET, de Wit M, Eder L, Fallon L, FitzGerald O, Gladman DD, Goel N, Holland R, Lindsay C, Maxwell L, Mease P, Orbai AM, Shea B, Strand V, Veale DJ, Tillett W, Ogdie A. Endorsement of the 66/68 Joint Count for the Measurement of Musculoskeletal Disease Activity: OMERACT 2018 Psoriatic Arthritis Workshop Report. J Rheumatol. 2019 Aug;46(8):996-1005. doi: 10.3899/jrheum.181089. Epub 2019 Feb 15. PMID 30770518
- [Background] Ramiro S, Nikiphorou E, Sepriano A, Ortolan A, Webers C, Baraliakos X, Landewe RBM, Van den Bosch FE, Boteva B, Bremander A, Carron P, Ciurea A, van Gaalen FA, Geher P, Gensler L, Hermann J, de Hooge M, Husakova M, Kiltz U, Lopez-Medina C, Machado PM, Marzo-Ortega H, Molto A, Navarro-Compan V, Nissen MJ, Pimentel-Santos FM, Poddubnyy D, Proft F, Rudwaleit M, Telkman M, Zhao SS, Ziade N, van der Heijde D. ASAS-EULAR recommendations for the management of axial spondyloarthritis: 2022 update. Ann Rheum Dis. 2023 Jan;82(1):19-34. doi: 10.1136/ard-2022-223296. Epub 2022 Oct 21. PMID 36270658
- [Background] Smolen JS, Landewe RBM, Bergstra SA, Kerschbaumer A, Sepriano A, Aletaha D, Caporali R, Edwards CJ, Hyrich KL, Pope JE, de Souza S, Stamm TA, Takeuchi T, Verschueren P, Winthrop KL, Balsa A, Bathon JM, Buch MH, Burmester GR, Buttgereit F, Cardiel MH, Chatzidionysiou K, Codreanu C, Cutolo M, den Broeder AA, El Aoufy K, Finckh A, Fonseca JE, Gottenberg JE, Haavardsholm EA, Iagnocco A, Lauper K, Li Z, McInnes IB, Mysler EF, Nash P, Poor G, Ristic GG, Rivellese F, Rubbert-Roth A, Schulze-Koops H, Stoilov N, Strangfeld A, van der Helm-van Mil A, van Duuren E, Vliet Vlieland TPM, Westhovens R, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2022 update. Ann Rheum Dis. 2023 Jan;82(1):3-18. doi: 10.1136/ard-2022-223356. Epub 2022 Nov 10. PMID 36357155
- [Background] Wolfe F, Clauw DJ, Fitzcharles MA, Goldenberg DL, Hauser W, Katz RL, Mease PJ, Russell AS, Russell IJ, Walitt B. 2016 Revisions to the 2010/2011 fibromyalgia diagnostic criteria. Semin Arthritis Rheum. 2016 Dec;46(3):319-329. doi: 10.1016/j.semarthrit.2016.08.012. Epub 2016 Aug 30. PMID 27916278
- [Background] SCORE2-OP working group and ESC Cardiovascular risk collaboration. SCORE2-OP risk prediction algorithms: estimating incident cardiovascular event risk in older persons in four geographical risk regions. Eur Heart J. 2021 Jul 1;42(25):2455-2467. doi: 10.1093/eurheartj/ehab312. PMID 34120185
- [Background] SCORE2 working group and ESC Cardiovascular risk collaboration. SCORE2 risk prediction algorithms: new models to estimate 10-year risk of cardiovascular disease in Europe. Eur Heart J. 2021 Jul 1;42(25):2439-2454. doi: 10.1093/eurheartj/ehab309. PMID 34120177
- [Background] Prevoo ML, van 't Hof MA, Kuper HH, van Leeuwen MA, van de Putte LB, van Riel PL. Modified disease activity scores that include twenty-eight-joint counts. Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. Arthritis Rheum. 1995 Jan;38(1):44-8. doi: 10.1002/art.1780380107. PMID 7818570
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Machado PM, Landewe R, Heijde DV; Assessment of SpondyloArthritis international Society (ASAS). Ankylosing Spondylitis Disease Activity Score (ASDAS): 2018 update of the nomenclature for disease activity states. Ann Rheum Dis. 2018 Oct;77(10):1539-1540. doi: 10.1136/annrheumdis-2018-213184. Epub 2018 Feb 16. No abstract available. PMID 29453216
- [Background] Naredo E, D'Agostino MA, Wakefield RJ, Moller I, Balint PV, Filippucci E, Iagnocco A, Karim Z, Terslev L, Bong DA, Garrido J, Martinez-Hernandez D, Bruyn GA; OMERACT Ultrasound Task Force*. Reliability of a consensus-based ultrasound score for tenosynovitis in rheumatoid arthritis. Ann Rheum Dis. 2013 Aug;72(8):1328-34. doi: 10.1136/annrheumdis-2012-202092. Epub 2012 Sep 14. PMID 22984169
- [Background] Zabotti A, Sakellariou G, Tinazzi I, Idolazzi L, Batticciotto A, Canzoni M, Carrara G, De Lucia O, Figus F, Girolimetto N, Macchioni P, McConnell R, Possemato N, Iagnocco A. Novel and reliable DACTylitis glObal Sonographic (DACTOS) score in psoriatic arthritis. Ann Rheum Dis. 2020 Aug;79(8):1037-1043. doi: 10.1136/annrheumdis-2020-217191. Epub 2020 May 19. PMID 32430315
- [Background] Balint PV, Terslev L, Aegerter P, Bruyn GAW, Chary-Valckenaere I, Gandjbakhch F, Iagnocco A, Jousse-Joulin S, Moller I, Naredo E, Schmidt WA, Wakefield RJ, D'Agostino MA; OMERACT Ultrasound Task Force members. Reliability of a consensus-based ultrasound definition and scoring for enthesitis in spondyloarthritis and psoriatic arthritis: an OMERACT US initiative. Ann Rheum Dis. 2018 Dec;77(12):1730-1735. doi: 10.1136/annrheumdis-2018-213609. Epub 2018 Aug 3. PMID 30076154
- [Background] D'Agostino MA, Terslev L, Aegerter P, Backhaus M, Balint P, Bruyn GA, Filippucci E, Grassi W, Iagnocco A, Jousse-Joulin S, Kane D, Naredo E, Schmidt W, Szkudlarek M, Conaghan PG, Wakefield RJ. Scoring ultrasound synovitis in rheumatoid arthritis: a EULAR-OMERACT ultrasound taskforce-Part 1: definition and development of a standardised, consensus-based scoring system. RMD Open. 2017 Jul 11;3(1):e000428. doi: 10.1136/rmdopen-2016-000428. eCollection 2017. PMID 28948983
- [Background] Schoels MM, Aletaha D, Alasti F, Smolen JS. Disease activity in psoriatic arthritis (PsA): defining remission and treatment success using the DAPSA score. Ann Rheum Dis. 2016 May;75(5):811-8. doi: 10.1136/annrheumdis-2015-207507. Epub 2015 Aug 12. PMID 26269398
- [Background] Rudwaleit M, van der Heijde D, Landewe R, Listing J, Akkoc N, Brandt J, Braun J, Chou CT, Collantes-Estevez E, Dougados M, Huang F, Gu J, Khan MA, Kirazli Y, Maksymowych WP, Mielants H, Sorensen IJ, Ozgocmen S, Roussou E, Valle-Onate R, Weber U, Wei J, Sieper J. The development of Assessment of SpondyloArthritis international Society classification criteria for axial spondyloarthritis (part II): validation and final selection. Ann Rheum Dis. 2009 Jun;68(6):777-83. doi: 10.1136/ard.2009.108233. Epub 2009 Mar 17. PMID 19297344
- [Background] Taylor W, Gladman D, Helliwell P, Marchesoni A, Mease P, Mielants H; CASPAR Study Group. Classification criteria for psoriatic arthritis: development of new criteria from a large international study. Arthritis Rheum. 2006 Aug;54(8):2665-73. doi: 10.1002/art.21972. PMID 16871531
- [Background] Mease P, Setty A, Papp K, Van den Bosch F, Tsuji S, Keiserman M, Carter K, Li Y, McCaskill R, McDearmon-Blondell E, Wung P, Tillett W. Upadacitinib in patients with psoriatic arthritis and inadequate response to biologics: 3-year results from the open-label extension of the randomised controlled phase 3 SELECT-PsA 2 study. Clin Exp Rheumatol. 2023 Nov;41(11):2286-2297. doi: 10.55563/clinexprheumatol/8l7bbk. Epub 2023 Jul 5. PMID 37404160
- [Background] McInnes IB, Kato K, Magrey M, Merola JF, Kishimoto M, Haaland D, Chen L, Duan Y, Liu J, Lippe R, Wung P. Efficacy and Safety of Upadacitinib in Patients with Psoriatic Arthritis: 2-Year Results from the Phase 3 SELECT-PsA 1 Study. Rheumatol Ther. 2023 Feb;10(1):275-292. doi: 10.1007/s40744-022-00499-w. Epub 2022 Oct 15. PMID 36243812
- [Background] Coates LC, Garrood T, Gullick N, Helliwell P, Kent T, Marks J, Tillett W, Kaur-Papadakis D, Tahir H, van Haaren S, McInnes I. Upadacitinib response rates in patients with psoriatic arthritis enrolled in the SELECT-PsA-1 and SELECT-PsA-2 trials assessed according to modified PsARC. Rheumatology (Oxford). 2022 Dec 23;62(1):e1-e3. doi: 10.1093/rheumatology/keac388. No abstract available. PMID 35799375
- [Background] Fleischmann R, Mysler E, Bessette L, Peterfy CG, Durez P, Tanaka Y, Swierkot J, Khan N, Bu X, Li Y, Song IH. Long-term safety and efficacy of upadacitinib or adalimumab in patients with rheumatoid arthritis: results through 3 years from the SELECT-COMPARE study. RMD Open. 2022 Feb;8(1):e002012. doi: 10.1136/rmdopen-2021-002012. PMID 35121639
- [Background] McInnes IB, Anderson JK, Magrey M, Merola JF, Liu Y, Kishimoto M, Jeka S, Pacheco-Tena C, Wang X, Chen L, Zueger P, Liu J, Pangan AL, Behrens F. Trial of Upadacitinib and Adalimumab for Psoriatic Arthritis. N Engl J Med. 2021 Apr 1;384(13):1227-1239. doi: 10.1056/NEJMoa2022516. PMID 33789011
- [Background] Coates LC, Corp N, van der Windt DA, O'Sullivan D, Soriano ER, Kavanaugh A. GRAPPA Treatment Recommendations: 2021 Update. J Rheumatol. 2022 Jun;49(6 Suppl 1):52-54. doi: 10.3899/jrheum.211331. Epub 2022 Mar 15. PMID 35293339
- [Background] Gossec L, Baraliakos X, Kerschbaumer A, de Wit M, McInnes I, Dougados M, Primdahl J, McGonagle DG, Aletaha D, Balanescu A, Balint PV, Bertheussen H, Boehncke WH, Burmester GR, Canete JD, Damjanov NS, Kragstrup TW, Kvien TK, Landewe RBM, Lories RJU, Marzo-Ortega H, Poddubnyy D, Rodrigues Manica SA, Schett G, Veale DJ, Van den Bosch FE, van der Heijde D, Smolen JS. EULAR recommendations for the management of psoriatic arthritis with pharmacological therapies: 2019 update. Ann Rheum Dis. 2020 Jun;79(6):700-712. doi: 10.1136/annrheumdis-2020-217159. PMID 32434812
- [Background] Celis R, Cuervo A, Ramirez J, Canete JD. Psoriatic Synovitis: Singularity and Potential Clinical Implications. Front Med (Lausanne). 2019 Feb 11;6:14. doi: 10.3389/fmed.2019.00014. eCollection 2019. PMID 30805340
- [Background] McGonagle D, Lories RJ, Tan AL, Benjamin M. The concept of a "synovio-entheseal complex" and its implications for understanding joint inflammation and damage in psoriatic arthritis and beyond. Arthritis Rheum. 2007 Aug;56(8):2482-91. doi: 10.1002/art.22758. No abstract available. PMID 17665450